CLINICAL TRIAL: NCT00627770
Title: Validation of a Procedure Using Bioimpedance to Measure the Edema of Lower Leg of Patients After Total Knee Surgery
Brief Title: Lower Leg Edema Evaluation After Total Knee Arthroplasty Using Bioimpedance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Claude Pichonnaz/ HES-professor and physiotherapist, HECVSanté (University of Applied Sciences in Health)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HECVSante01; SAGE-X 19860
Record Dates: First submitted 2008-02-06; First posted 2008-03-03 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Edema
Keywords: Physical Therapy - Therapeutics - Edema; Arthroplasty replacement knee; Treatment outcome
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: bioimpedance spectroscopy ImpediMed SFB7 Brisbane Australia — edema evaluation using bioimpedance

SUMMARY:
The purpose of this study is to evaluate the applicability and measurement properties of bioimpedance spectroscopy for postsurgical edema assessment after total knee arthroplasty

DETAILED DESCRIPTION:
Current measurement techniques of edema are not adapted or not convenient for assessment in the post surgical environment. Developement of a convenient, quick and reliable method could be useful to facilitate edema evaluation in this context.

ELIGIBILITY:
Inclusion Criteria:

* knee replacement surgery

Exclusion Criteria:

* pacemaker
* cardiac defibrillator
* other metallic implant than knee arthroplasty

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
bioimpedance ratio right/left | presurgery, 2 and 8 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claude A Pichonnaz, physiother., Principal Investigator — Haute Ecole de Santé Vaud; Brigitte M Jolles, PhD MER MSc, Study Director — Département de l'Appareil Locomoteur - CHUV + Faculté des sciences et techniques de l'ingénieur (STI) - EPFL; Correvon Marc, Engineer, Principal Investigator — Haute Ecole Vaudoise d'Ingénierie et de Gestion
Locations (1):
- Département de l'Appareil Locomoteur - CHUV, Lausanne, Switzerland

REFERENCES:
- [Derived] Pichonnaz C, Bassin JP, Lecureux E, Currat D, Jolles BM. Bioimpedance spectroscopy for swelling evaluation following total knee arthroplasty: a validation study. BMC Musculoskelet Disord. 2015 Apr 25;16:100. doi: 10.1186/s12891-015-0559-5. PMID 25907994